CLINICAL TRIAL: NCT03526302
Title: Register About Change of hsTROPoninT After Implantation of a Subcutaneous Implantable Cardioverter-Defibrillator
Brief Title: TroponinT After Subcutaneous Cardioverter-Defibrillator Implantation
Acronym: TROPIC
Status: Completed | Type: Observational
Sponsor: Deutsches Herzzentrum Muenchen (Other)
Responsible Party: Sponsor
Other Study IDs: GER-EP-018
Record Dates: First submitted 2018-05-03; First posted 2018-05-16 (Actual); Last update posted 2023-03-20 (Actual); Status verified 2023-03

CONDITIONS: Sudden Cardiac Death
MeSH Terms: conditions — Death, Sudden, Cardiac

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Serum Troponin levels pre- and postoperatively will be compared in patients receiving an entirely subcutaneous cardioverter-defibrillator.

DETAILED DESCRIPTION:
To analyze the periprocedural myocardial damage the pre- and postoperative assessment of serum levels of high sensitive TroponinT (hsTnT) is done. The main objectives of the TROPIC register are to evaluate the level of high sensitive TroponinT before and after S-ICD device implantation and to compare these changes in TroponinT-levels with those after standard transvenous ICD-implantation.

ELIGIBILITY:
Inclusion Criteria:

* Indication for the implantation of an entirely subcutaneous cardioverter-defibrillator

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with the indication for the implantation of an entirely subcutaneous cardioverter-defibrillator
Sampling Method: Non-Probability Sample
Enrollment: 43 (Actual)
Dates: Start 2018-04-01 (Actual); Primary Completion 2020-09-30 (Actual); Study Completion 2020-09-30 (Actual)

PRIMARY OUTCOMES:
High sensitive TroponinT | 24 hours
  Difference between pre- and postoperative high sensitive TroponinT serum levels

CONTACTS AND LOCATIONS:
Overall Officials: Christof Kolb, MD, Principal Investigator — Deutsches Herzzentrum München
Locations (1):
- Deutsches Herzzentrum München, München, Germany

REFERENCES:
- [Result] Weigand S, O'Connor M, Blazek P, Kantenwein V, Friedrich L, Grebmer C, Schaarschmidt C, von Olshausen G, Reents T, Deisenhofer I, Lennerz C, Kolb C. Release of high-sensitive TROPonin T by implantation of an entirely subcutaneous Implantable Cardioverter-defibrillator compared to a conventional transvenous approach: the TROPIC registry. J Interv Card Electrophysiol. 2021 Oct;62(1):75-81. doi: 10.1007/s10840-020-00874-z. Epub 2020 Sep 21. PMID 32959177